CLINICAL TRIAL: NCT04387266
Title: A Retrospective Real-world Study in Patients With Nasopharyngeal Carcinoma: to Evaluate the Efficacy and Feasibility of Modified Reduce-volume Target IMRT in the Treatment of Patients With Non-metastatic NPC
Brief Title: To Evaluate the Efficacy and Feasibility of Modified Reduce-volume Target IMRT in the Treatment of Patients With Non-metastatic NPC
Status: Completed | Type: Observational
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: NPC004
Record Dates: First submitted 2020-05-10; First posted 2020-05-13 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Modified reduce-volume target IMRT: Patients with newly diagnosed, non-metastatic NPC was given modified reduce-volume target IMRT
  Interventions: Radiation: modified reduce-volume target IMRT

INTERVENTIONS:
Radiation: modified reduce-volume target IMRT — The gross tumor volume of the nasopharynx and neck nodes (GTVnx and GTVnd) were delineated according to the tumor extension. The CTVnx was defined as GTVnx + nasopharynx mucosa + 8mm +corresponding anatomical structure without the delineation of CTV1. The CTVnd was defined as GTVnd plus the elective neck area. The prescribe doses of GTVnx/GTVnd, CTVnx, CTVnd were 66-70Gy,54-56Gy and 50-54Gy in 31-35 fractions, respectively.

SUMMARY:
This is a retrospective real-world study to evaluate the efficacy and feasibility of modified reduce-volume target IMRT in the treatment of patients with non-metastatic NPC

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis (pathologically confirmed by nasopharyngeal biopsy) was nasopharyngeal carcinoma;
2. Newly diagnosed, non-metastatic and treated with modified reduce-volume IMRT;
3. Patients with baseline MRI date of nasopharynx and neck, and completed the first course of treatment in our hospital;
4. Diagnosis time: November 1, 2014 to December 31 , 2017

Exclusion Criteria:

1. Disease progression during IMRT;
2. Previous malignancy or other concomitant malignant diseases;
3. The evaluation information of tumor efficacy can not be obtained;
4. Receive blind treatment in other clinical research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-metastatic NPC patients treated with modified reduce-volume target IMRT in our institution
Sampling Method: Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Local failure-free survival (LFFS) | 60 month
  The duration of time to LFFS was calculated from the date of histological diagnosis until documented treatment local failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of radiation oncology, Fujian cancer hospital, Fuzhou, Fujian, China